CLINICAL TRIAL: NCT04590872
Title: A Pilot Study to Evaluate the Safety and Feasibility of Autologous Tolerogenic Dendritic Cells Loaded With Proinsulin Peptide (C19-A3) in Patients With Type 1 Diabetes
Brief Title: An Immunotherapy Vaccine (PIpepTolDC) for the Treatment of Patients With Type 1 Diabetes
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18279
Record Dates: First submitted 2020-10-06; First posted 2020-10-19 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Autologous Tolerogenic Dendritic Cell with Proinsulin Peptide (PIpepTolDC) (Experimental): After completion of leukapheresis, patients receive a prime dose of PIpepTolDC intradermally (ID) on Day 0, followed by a boost dose of PIpepTolDC ID on Day 28.
  Interventions: Biological: Tolerogenic Dendritic Cell Vaccine

INTERVENTIONS:
Biological: Tolerogenic Dendritic Cell Vaccine — PIpepTolDCs

SUMMARY:
This phase I trial investigates the side effects of PIpepTolDC vaccine in treating patients with type 1 diabetes who use insulin and don't have any other diabetes-related health complications. Type 1 diabetes is an autoimmune disease. This means that the immune system, which usually protects against foreign invaders like bacteria and viruses, attacks the body's insulin-producing betacells in the pancreas (autoimmune response). Overtime, the beta cells are destroyed by the immune system. To stay alive, people with type 1 diabetes must use insulin. PIpepTolDC vaccine is a type of immunotherapy (a treatment that uses a person's own immune system) that works like an allergy shot. The vaccine is made using one's own immune cells (dendritic cells) and a beta cell protein. The vaccine may teach the immune system to stop attacking the beta cells, which may help the beta cells recover and make enough insulin to control blood sugar levels. The vaccine may also help reduce future type 1 diabetes related complications.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to undergo leukapheresis
* Willingness to be followed for about 2 years post-prime dose
* For participants who have a personal continuous glucose monitoring device (CGMD): Willingness to wear a second CGMD during mandated study CGMD visits
* Diagnosis of type 1 diabetes based on American Diabetes Association (ADA) criteria
* Historical presence of at least one type-1 diabetes associated autoantibody

  * GAD specific autoantibodies (glutamic acid decarboxylase autoantibodies [GADA])
  * Islet cell cytoplasmic autoantibodies (ICA)
  * Islet-antigen 2 specific autoantibody (IA-2A)
  * Zinc transporter 8 specific autoantibody (ZNT8A); and/or
  * Insulin autoantibody (IAA) (must have been obtained within 7 days of initiating exogenous insulin replacement therapy)
* Time from diagnosis to screening mixed meal tolerance test (MMTT) must be >= 1 year but =< 4 years
* Stable glycemic control per participant's physician
* HbA1c =< 7.5% (=< 58 mmol/mol)
* Non-fasting C-peptide > 0.017 nmol/L
* Stimulated peak C-peptide levels > 0.2 nmol/L from a 2-hour screening MMTT
* Positive for *04:01 allele, *04:02 allele and/or *04:04 allele at the human leukocyte antigen (HLA)-DRB1 gene locus
* Does not possess the protective HLA-DRB1*15:01-DQA1*01:02-DQB1*06:02 haplotype
* Adequate self-assessment of blood glucose values and recording of glucose values, and administered insulin doses as deemed sufficient by the participant's physician
* No diagnosis of type 1 diabetes related microvascular/macrovascular complications (e.g. nephropathy, retinopathy and neuropathy)
* Deemed acceptable for autologous cell collection (i.e. leukapheresis)
* Only for those who are naive to CGMD use: Deemed able to correctly use a CGM device following training session with a certified diabetes educator and manufacturer representative
* Must meet organ function criteria

Exclusion Criteria:

* Other investigational agents, biologics
* Anti-inflammatory therapy

  * Exception: Over-the-counter (OTC) anti-inflammatory agents (e.g. ibuprofen, Tylenol) are generally allowed. However, those requiring chronic OTC anti-inflammatory agents and unable to stop during mandated CGMD study visits will be excluded
* Systemic corticosteroids within 28 days prior to leukapheresis
* Systemic immunosuppressive therapy (e.g. cyclosporine-A, cyclophosphamide)
* Monoclonal antibody therapy
* Allergen immunotherapy within 28 days prior to leukapheresis
* Vaccine(s) within 28 days prior to leukapheresis
* Prior allogeneic organ transplant
* Beta-cell stimulants (e.g. sulfonylureas such as glimepiride), glucagon-like peptide-1 agonists, dipeptidyl peptidase-IV inhibitors (exception: Those with acute exposure to these agents during T1D misdiagnosis may be permitted per PI discretion)
* Insulin sensitizers (e.g. metformin, thiazolidinediones) within 2 months of leukapheresis
* History of insulin sensitizer use (e.g. metformin, thiazolidinediones) ≥ 2 months
* Other autoimmune/inflammatory disorders (exceptions: (i) Type 1 diabetes. (ii) Asymptomatic patients with incidental autoantibody titres may be permitted per PI discretion)
* Other autoimmune/inflammatory disorders (exception type 1 diabetes)
* Active infection requiring antibiotics and/or anti-virals
* Known history of HIV, HBV, HCV, HTLV, syphilis
* History of positive purified protein derivative (PPD) skin test
* History of atopy requiring systemic treatment and/or history of severe allergic reactions
* History or current malignancy
* Unstable cardiac disease
* History of vascular disease (e.g. deep vein thrombosis, stroke)
* Clinically significant uncontrolled illness
* Females only: pregnant or breastfeeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 2 years
  Toxicity and adverse events (except hypoglycemia and diabetic ketoacidosis [DKA]) will be recorded using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. Hypoglycemia events and DKA will be defined per American Diabetes Association (ADA) grading systems.Observed toxicities will be summarized by type, severity (by CTCAE v 5.0 and nadir or maximum values for lab measures), date of onset, duration, reversibility, and attribution.
Apheresis duration | up to 2 years
  Measured in hours.
Number of CD14+ monocytes | up to 2 years
  Number of CD14+ monocytes collected during apheresis
TolDC recovery after culture | up to 2 years
  Number of TolDC generated from CD14+ monocytes
Number of successful manufactured products | Up to 2 years
  Number of manufactured products that meet the required cell dose/day, sterility (e.g. endotoxin and gram staining), and viability compared to the total number of products manufactured.

SECONDARY OUTCOMES:
Change in stimulated C-peptide area under the curve | Baseline up to 2 years of follow up
  Assessed via 2-hr mixed meal tolerance test (MMTT). C-peptide preservation is defined as the maintenance of baseline C-peptide levels.
Change in interferon (IFN)-gamma and IL-10 producing CD4+ T cells | Baseline up to 2 years of follow up
  Will be assessed in response to pro-insulin peptide C19-A3, and assessed via cytokine enzyme-linked immunosorbent spot assay.
Change in T cell responsiveness | Baseline up to 2 years of follow up
  Will assess for changes in T cell responsiveness to pro-insulin peptide C19-A3 compared to other antigens. Assessed via Lymphocyte Simulation Test.
Change in the number of CD8+ autoreactive T cells | Baseline up to 2 years of follow up
  Assessed via quantum dot (Q-DOT) nanotechnology assay.
Change in immune phenotype | Baseline up to 2 years of follow up
  Will analyze for changes in immune cell populations via flow cytometry
Change in islet autoantibodies | Baseline up to 2 years of follow up
  Will analyze for changes in IAA, GAA, IA-2A, ZnT8A via enzyme-linked immunosorbent assay.
Change in glycosylated hemoglobin A1c (HbA1c) levels | Baseline up to 2 years of follow up
  HbA1c levels will be assessed via blood test
Change in exogenous insulin use (units/kg) | Baseline up to 2 years of follow up
  Insulin usage will be recorded daily from the insulin pump and/or participant insulin use logs. The mean daily insulin usage over the 10 consecutive days (IU units/kg body weight/day) preceding the clinic visit will be calculated for each participant.
Change in blood glucose levels | Baseline up to 2 years of follow up
  Will include clinically important/severe hypoglycemia, hyperglycemia and DKA events as assessed by ADA grading systems. Levels of glucose will be assessed from bloods samples taken during the MMTT and from insulin pump/participant insulin logs

CONTACTS AND LOCATIONS:
Overall Officials: Behrouz Salehian-Dardashti, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States